CLINICAL TRIAL: NCT01452529
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study With an Open-label Run-in to Assess the Efficacy and Safety of Hydrocodone Bitartrate (HYD) Tablets 20 to 120 mg Once-daily in Subjects With Moderate to Severe Chronic Low Back Pain
Brief Title: Efficacy and Safety of Hydrocodone Bitartrate (HYD) in Subjects With Moderate to Severe Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HYD3002
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Chronic Low Back Pain
Keywords: Pain; Opioid
MeSH Terms: conditions — Pain | interventions — Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrocodone bitartrate (Experimental): Hydrocodone bitartrate (HYD) once daily (q24h) tablets
  Interventions: Drug: Hydrocodone bitartrate q24h film-coated tablets
- Placebo (Placebo Comparator): Placebo to match hydrocodone bitartrate once daily tablets
  Interventions: Drug: Placebo to match hydrocodone bitartrate q24h tablets

INTERVENTIONS:
Drug: Hydrocodone bitartrate q24h film-coated tablets — Hydrocodone bitartrate q24h film-coated tablets 20 - 120 mg once daily
  Other Names: Hysingla ER
  Arms: Hydrocodone bitartrate
Drug: Placebo to match hydrocodone bitartrate q24h tablets — Placebo to match hydrocodone bitartrate q24h film coated tablets 20 - 120 mg once daily
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy and safety of HYD tablets 20 to 120 mg once-daily dose compared to placebo in subjects with moderate to severe chronic low back pain uncontrolled by their current stable analgesic regimen

ELIGIBILITY:
Inclusion Criteria include:

* Male and female subjects ≥ 18 years of age with moderate to severe, chronic low back pain (lasting several hours daily) as their predominant pain condition for at least 3 months prior to the screening visit;
* Subjects whose low back pain is not adequately treated prior to the screening visit with their stable incoming analgesic regimen;
* Subjects deemed by the investigator/medically qualified designee (must be MD or DO) to be appropriate candidates for the protocol specified, around the clock HYD therapeutic regimen;
* Female subjects who are premenopausal or postmenopausal less than 1 year and who have not had surgical sterilization (ie, tubal ligation, partial or complete hysterectomy) must have a negative serum pregnancy test, be nonlactating, and willing to use adequate and reliable contraception throughout the study (eg, barrier with additional spermicidal foam or jelly, intra-uterine device, hormonal contraception).

Exclusion Criteria include:

* Subjects taking > 100 mg/day oxycodone or equivalent during last 14 days prior to screening visit;
* Subjects who cannot or will not agree to completely stop all incoming opioid and nonopioid analgesic medications and other medications used for chronic pain, excluding herbal and nutraceutical medications;
* Subjects who cannot or will not agree to stop local regional pain treatments during the study (nerve/plexus blocks or ablation, neurosurgical procedures for pain control, botulinum toxin injections for control of chronic low back pain, steroid injections in the lower back or inhalation analgesia). The subject must not have had a nerve/plexus block within 4 weeks of the screening visit, neuroablation within 6 months of the screening visit, a botulinum toxin injection in the low back region within 3 months of the screening visit, steroid injections in the lower back within 6 weeks of the screening visit, or intravenous or intramuscular steroid injections within 4 weeks of the screening visit;
* Subjects who have used any investigational medication within 30 days prior to the first dose of study medication;
* Subjects with any history of seizures (subjects with history of pediatric febrile seizures may participate in the study) or increase in intracranial pressure;
* Subjects with current uncontrolled depression or other uncontrolled psychiatric disorder (subjects with controlled depression or other psychiatric disorder must be on a stable medication for ≥ 1 month prior to the screening visit to participate in the study);
* Subjects with a history of alcohol, medication, or illicit drug abuse or addiction and/or history of opioid abuse or addiction at any time;
* Subjects with clinically unstable cardiac disease, including: unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or indwelling pacemaker;
* Subjects with unstable respiratory disease that, in the opinion of the investigator, precludes entry into this study;
* Subjects with evidence of impaired liver function upon entry into the study (laboratory test values ≥ 3 times the upper limit of the laboratory reference (normal) range (ULN) for aspartate transaminase [AST/SGOT] or alanine transaminase [ALT/SGPT], or values > 2 times the ULN for alkaline phosphatase), or total bilirubin level > 1.5 times the ULN or, in the opinion of the investigator/medically qualified designee (must be MD or DO), liver function impairment to the extent that the subject should not participate in this study;
* Subjects with evidence of impaired kidney function upon entry into the study (ie, serum creatinine ≥ 2.5 mg/dL);
* Subjects with biliary tract disease, hypothyroidism, adrenal cortical insufficiency, or any other medical condition that, in the opinion of the investigator, is inadequately treated and precludes entry into the study;
* Subjects who had surgical procedures directed towards the source of chronic low back pain within 6 months of the screening visit or scheduled for surgery of the lower back or any other major surgery during the study conduct period;
* Subjects with history of malignancy within past 2 years, with exception of basal cell carcinoma that has been successfully treated;
* Subjects with any condition in which opioids are contraindicated, eg, severe respiratory depression with hypoxia and/or hypercapnia, severe chronic obstructive lung disease, cor pulmonale, severe bronchial asthma, or paralytic ileus;
* Subjects who are allergic to hydrocodone or who have a history of allergies to other opioids. This does not include subjects who have experienced common opioid side effects (eg, nausea, constipation);
* Subjects receiving monoamine oxidase inhibitors (MAOIs) or who have been taking MAOIs within 2 weeks of the screening visit.

Other protocol-specific inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (102):
  - Alliance Clinical Research, Birmingham, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Redpoint Research, Phoenix, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Redpoint Research, Tucson, Arizona
  - ACRI-Phase 1, LLC, Anaheim, California
  - Orange County Research Institute, Anaheim, California
  - United Clinical Research Center, Inc., Anaheim, California
  - Research Center of Fresno, Inc., Fresno, California
  - TriWest Research Associates, La Mesa, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Skyline Research, LLC, Long Beach, California
  - Center for Clinical Research, Inc., Richmond, California
  - Northern California Research, Sacramento, California
  - Encompass Clinical Research, Spring Valley, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Meridien Research, Bradenton, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Florida Health Center, Fort Lauderdale, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Fidelity Clinical Research, Inc., Lauderhill, Florida
  - Neuroscience Consultants LLC, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Journey Research, Inc, Oldsmar, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - Peninsula Research Inc., Ormond Beach, Florida
  - Advent Clinical Research Centers, Inc., Pinellas Park, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Sarasota Research, LLC, Sarasota, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Southeast Regional Research Group, Columbus, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Taylor Research, LLC, Marietta, Georgia
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Atlanta Knee and Shoulder Clinic, PC, Stockbridge, Georgia
  - Illinois Center for Clinical Research, Chicago, Illinois
  - Rehabilitation Associates of Indiana, Indianapolis, Indiana
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - ICRI, Overland Park, Kansas
  - Community Research, Crestview Hills, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - IRC Clinics, Inc., Towson, Maryland
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - QUEST Research Institute, Bingham Farms, Michigan
  - Medical Research Associates, Inc., Traverse City, Michigan
  - Healthcare Research Network, Hazelwood, Missouri
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Advance Clinical Research, St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Research Facility, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - CRI Worldwide LLC, Willingboro, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - The Medical Research Network, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - PMG Research of Wilmington LLC, Wilmington, North Carolina
  - Clinical Trials of America, Inc., Winston-Salem, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Daystar Clinical Research, Inc., Akron, Ohio
  - IVA Research, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Bone Joint and Spine Surgeons, Inc., Toledo, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Allegheny Pain Management, P.C., Altoona, Pennsylvania
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Founders Research Corporation, Philadelphia, Pennsylvania
  - Tipton Medical & Diagnostic Center, Tipton, Pennsylvania
  - Hartwell Research Group, Anderson, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Comprehensive Pain Specialists, LLC, Hendersonville, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Heartland Medical, PC, New Tazewell, Tennessee
  - HCCA Clinical Research Solutions, Smyrna, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - Heights Doctor's Clinic, Houston, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Sun Research Institute, San Antonio, Texas
  - Aspen Clinical Research, Orem, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - HypotheTest, LLC, Roanoke, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Washington Center for Pain Management, Edmonds, Washington

REFERENCES:
- [Result] Wen W, Sitar S, Lynch SY, He E, Ripa SR. A multicenter, randomized, double-blind, placebo-controlled trial to assess the efficacy and safety of single-entity, once-daily hydrocodone tablets in patients with uncontrolled moderate to severe chronic low back pain. Expert Opin Pharmacother. 2015;16(11):1593-606. doi: 10.1517/14656566.2015.1060221. Epub 2015 Jun 26. PMID 26111544
- [Derived] Campbell K, Kutz JW Jr, Shoup A, Wen W, Lynch SY, He E, Ripa SR. Evaluation of the Ototoxicity Potential of Once-Daily, Single-Entity Hydrocodone in Patients with Chronic Pain: Results of Two Phase-3 Clinical Studies. Pain Physician. 2017 Jan-Feb;20(1):E183-E193. PMID 28072811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject first visit: 23-March-2012; Last subject last visit: 03-September-2013. The study was conducted at medical/research sites in the United States.
Pre-assignment Details: Subjects with moderate to severe chronic low back pain uncontrolled by their current stable analgesic regimen were included.
Groups:
- Open-label Run-in Dose-titration Period Hydrocodone Bitartrate: The open-label run-in dose-titration period was designed to assess subjects qualification for randomization
Period: Run-in Period
Arm/Group | Open-label Run-in Dose-titration Period Hydrocodone Bitartrate | Hydrocodone Bitartrate | Placebo
Started | 905 | 0 | 0
Completed | 592 | 0 | 0
Not Completed | 313 | 0 | 0
Not completed — Adverse Event | 96 | 0 | 0
Not completed — Withdrawal by Subject | 49 | 0 | 0
Not completed — Lost to Follow-up | 19 | 0 | 0
Not completed — Lack of Efficacy | 46 | 0 | 0
Not completed — Confirmed or suspected diversion | 23 | 0 | 0
Not completed — Administrative | 21 | 0 | 0
Not completed — Did not qualify for Double-Blind Phase | 59 | 0 | 0
Period: Double-blind (DB) Period
Arm/Group | Open-label Run-in Dose-titration Period Hydrocodone Bitartrate | Hydrocodone Bitartrate | Placebo
Started | 0 | 296 (Four subjects were randomized but did not receive DB medication) | 292
Completed | 0 | 229 (4 subjects who did not receive DB medication were still counted as discontinued in the DB period) | 210
Not Completed | 0 | 67 | 82
Not completed — Adverse Event | 0 | 18 | 11
Not completed — Withdrawal by Subject | 0 | 15 | 14
Not completed — Lost to Follow-up | 0 | 5 | 3
Not completed — Lack of Efficacy | 0 | 16 | 44
Not completed — Confirmed or suspected diversion | 0 | 2 | 3
Not completed — Administrative | 0 | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocodone Bitartrate | Placebo | Total
Number analyzed (Participants) | 296 | 292 | 588
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (13.51) | 47.9 (13.23) | 48.6 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 166 | 338
  Male | 124 | 126 | 250
Race/Ethnicity, Customized [Number; unit: participants]
  White | 195 | 207 | 402
  Black or African American | 67 | 51 | 118
  Asian | 25 | 29 | 54
  American Indian or Alaska Native | 2 | 1 | 3
  Other | 7 | 4 | 11
Screening Baseline Pain Over the Last 24 Hours [Mean (Standard Deviation); unit: units on a scale] — "Average pain over the last 24 hours" score (on an 11-point numerical rating scale where 0 = no pain and 10 = pain as bad as you can imagine).
  units on a scale | 7.4 (1.13) | 7.4 (1.19) | 7.4 (1.16)

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Intensity for "Average Pain Over the Last 24 Hours" Score
Description: Mean pain intensity for "average pain over the last 24 hours" score (on an 11-point numerical rating scale where 0 = no pain and 10 = pain as bad as you can imagine).
Time Frame: Week 12
Population: The full analysis population (N = 588) was the group of subjects who were randomized and received at least 1 dose of double-blind study drug
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hydrocodone Bitartrate | Placebo
Number analyzed (Participants) | 296 | 292
units on a scale | 3.7 (0.13) | 4.2 (0.13)

2. Secondary Outcome: Medical Outcome Study Sleep Scale - Revised (MOS Sleep-R) - Sleep Disturbance Subscale
Description: The MOS Sleep-R is a brief, self-administered 12-item assessment designed to measure key aspects of sleep. It includes a sleep problems index and 6 subscales - sleep disturbance, sleep adequacy, daytime somnolence, snoring, awaken short of breath or with headache, and quantity of sleep. The sleep disturbance subscale comprised the responses to questions 1, 3, 7, and 8 on the assessment. The individual responses for each question were recorded on a 5-point scale with options ranging from 1 - "all of the time" to 5 - "none of the time". Sleep disturbance scores were transformed linearly on a scale of 0-100. A higher value indicates a better score; therefore, a higher score indicates a better sleep pattern.
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydrocodone Bitartrate | Placebo
Number analyzed (Participants) | 296 | 292
units on a scale
  Screening | 44.38 (9.262) | 44.72 (9.871)
  Week 4 | 50.38 (8.851) | 50.51 (9.156)
  Week 8 | 50.16 (8.879) | 51.16 (8.781)
  Week 12 | 51.57 (8.576) | 52.12 (8.779)

3. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC is an ordinal scale which assesses the change in overall status relative to the start of the study. The scale has only 1 item, which measures global change of overall status by the subject on a 7-point scale (very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse), where 1 = very much improved and 7 = very much worse. The proportion of subjects responding "very much improved" and "much improved" was summarized by treatment group.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Hydrocodone Bitartrate | Placebo
Number analyzed (Participants) | 296 | 292
Participants
  Total Subjects Completing PGIC | 283 | 267
  Subjects Responding Very Much or Much Improved | 173 | 130

4. Secondary Outcome: Responder Analysis for Subjects With a ≥ 30% Reduction in Pain Compared to Baseline
Description: A subject's response to treatment was defined as the percentage reduction from the screening mean pain score to the mean pain intensity at week 12 of the double-blind period.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Hydrocodone Bitartrate | Placebo
Number analyzed (Participants) | 296 | 292
Participants
  Number of Subjects Responding | 285 | 280
  Number of Subjects with ≥ 30% Reduction in Pain | 184 | 147

5. Secondary Outcome: Responder Analysis for Subjects With a ≥ 50% Reduction in Pain Compared to Baseline
Description: as for outcome 4
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Hydrocodone Bitartrate | Placebo
Number analyzed (Participants) | 296 | 292
Participants
  Number of Subjects Responding | 285 | 280
  Number of Subjects with ≥ 50% Reduction in Pain | 137 | 109

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from start of study participation through the period beyond study completion.
Description: AEs were learned of through spontaneous reports and/or subject interview, or were observed during physical examinations or other safety assessments. Ongoing AEs were followed until resolution or 30 days after last study drug dose. Serious AEs up to 30 days following the last study visit were followed until the AE or sequelae resolved or stabilized.
Groups:
- Open-label Run-in Dose-titration Period Hydrocodone Bitartrate: The open-label run-in dose-titration period was designed to assess subjects' qualification for randomization
Arm/Group | Open-label Run-in Dose-titration Period Hydrocodone Bitartrate | Hydrocodone Bitartrate | Placebo
Serious Adverse Events (participants affected / at risk) | 7/905 | 2/296 | 4/292
Other Adverse Events (participants affected / at risk) | 265/905 | 52/296 | 30/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Run-in Dose-titration Period Hydrocodone Bitartrate (N=905) | Hydrocodone Bitartrate (N=296) | Placebo (N=292)
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — Outcome: Death
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0 — Outcome: Death
Drug abuse (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Run-in Dose-titration Period Hydrocodone Bitartrate (N=905) | Hydrocodone Bitartrate (N=296) | Placebo (N=292)
Nausea (Gastrointestinal disorders) | 144 | 24 | 16
Constipation (Gastrointestinal disorders) | 85 | 10 | 7
Vomiting (Gastrointestinal disorders) | 65 | 18 | 9
Dizziness (Nervous system disorders) | 64 | 9 | 5
Headache (Nervous system disorders) | 59 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days